CLINICAL TRIAL: NCT04995224
Title: Psychophysiological and Biological Profiling of Chronic Pain in Patients With Inflammatory Bowel Disease
Brief Title: Mechanism of Chronic Pain in Patients With IBD
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Birmingham (Other); University of Cambridge (Other); Barking, Havering and Redbridge University Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); University College London Hospitals (Other); Royal Free Hospital NHS Foundation Trust (Other); King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 279414
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel diseases, IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — blood, stool samples, and colon biopsies from a maximum of 150 patients in study 1A
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Study 1A: Prospective cohort study with 150 newly diagnosed patients with inflammatory bowel disease
  Interventions: Other: Assessment of Psychophysiological factors; Biological: Assessment of Biological factors; Genetic: Assessment of Genetics; Behavioral: Assessment of Quality of Life
- Study 1B: Prospective cohort study with 450 newly diagnosed patients with IBD
  Interventions: Other: Assessment of Psychophysiological factors; Genetic: Assessment of Genetics; Behavioral: Assessment of Quality of Life; Biological: Assessment of Biological factors
- Study 2: Cross-sectional study with 10,000 patients in IBD Boost study
  Interventions: Other: Assessment of Psychophysiological factors; Genetic: Assessment of Genetics; Behavioral: Assessment of Quality of Life
- Study 3: Cross-sectional study with 15,000 patients in IBD BioResource
  Interventions: Other: Assessment of Psychophysiological factors; Genetic: Assessment of Genetics; Behavioral: Assessment of Quality of Life

INTERVENTIONS:
Other: Assessment of Psychophysiological factors — Investigating the presence of psychophysiological factors (depression, anxiety, catastrophizing) by questionnaires.
Biological: Assessment of Biological factors — Investigating autonomic nervous function using heart rate recording, colon biopsy samples, microbiota, and blood cytokines levels. (Colon biopsy samples are obtained when colonoscopy is performed for clinical reasons. Blood samples and stool samples will be taken when participants come to the hospital for colonoscopy)
  Groups: Study 1A
Genetic: Assessment of Genetics — Genetic data investigated by another cohort study (IBD BioResource study) will be utilized in the analysis of this study.
Behavioral: Assessment of Quality of Life — Investigating QOL by questionnaires.
Biological: Assessment of Biological factors — Investigating colon biopsy samples (Colon biopsy samples are obtained when colonoscopy is performed for clinical reasons).
  Groups: Study 1B

SUMMARY:
Abdominal pain is a common symptom in patients with inflammatory bowel disease (IBD). Up to 70 % of IBD patients experience pain when the disease is active. Even when patients with IBD are in remission, 20-50 % experience ongoing pain. The precise mechanism of developing chronic abdominal pain in patients with IBD in remission remains unknown.

The aim of this study is to identify psychophysiological and biological risk factors for the development of chronic abdominal pain in patients with newly diagnosed IBD (ulcerative colitis and Crohn's disease).

This study consists of 4 sections (Study 1A, 1B, 2, and 3):

Study 1A: We perform a longitudinal study in 150 patients with new-onset IBD over 18 months to identify risk factors related to the brain-gut axis for the development of chronic pain. This is a collaborative study with IBD BioResourse Inception study. We administer online questionnaires, collect stool and blood samples, and record heart rate. Other physiological data collected by the Inception study will be also used for the analysis.

Study 1B: This is also a collaborative study with the Inception study. We will apply for our detailed questionnaires for 7 days (as per study 1A) to be administered to all the new patients (n=450) that are included in the Inception study on a voluntary basis. Patients will be followed for 12 months.

Study 2 and 3: Study 2 and 3 are a questionnaire-based cross-sectional study in patients with IBD. The participants for study 2 are patients registered in IBD BOOST study and those for study 3 are patients registered in IBD BioResource (but not in IBD Boost study). Detailed online questionnaires will be administered to them. These studies are just one-day assessment.

DETAILED DESCRIPTION:
This study consists of 4 sections (Study 1A, 1B, 2, and 3).

Study 1A: We perform a longitudinal study in 150 patients with new-onset IBD (UC and CD) over 18 months to identify risk factors related to the brain-gut axis for the development of chronic pain.

First assessment period: On the first day of the study, we will have a video chat with the participant using one of the telecommunications applications (e.g. skype, zoom, Microsoft team, etc.) and obtain an electric consent form using DocuSign (https://www.docusign.co.uk/). Then, participants will be trained on how to use online validated questionnaires to evaluate their disease activity, symptoms and psychological state, presence or absence of irritable bowel syndrome (IBS), or pain elsewhere. Then, they will be asked to download a mobile phone camera heart rate variability app and be trained to use it. They will also be trained to use the experience sampling method (ESM) to profile gut symptoms and lifestyle via a smartphone app at 10 random times in a day.

After training, participants will fill out baseline online questionnaires using REDCap. Participants will also start answering questionnaires by ESM for 7 days and recording their heart rate (5 minutes) using the app once a day in the morning for 7 days.

2nd-4th assessment periods: Further assessment periods will be scheduled every 6 months. One-two days before each study period begins, we will remind the participants by email or phone call. On day 1, participants fill out the same online questionnaires (except personality, which is a stable trait) followed by 7 days ESM profiling as during their first assessment period. They will also be asked to record heart rate (5 minutes) once a day in the morning for 7days. Each patient will be followed at least 18 months until the 4th assessment period ends.

If patients agree, we will add online questionnaires to patients beyond the life of the grant (at 24 months and 36 months) when they are followed by the IBD BioResource inception study. (ESM and sample collection are not performed after 18 months follow)

This is a collaborative study with the IBD BioResource Inception study. The participants in our study will be asked to participate in the IBD BioResource Inception study as well. Biological data obtained by the BioResource Inception study, which will be used for the analysis.

Study 1B: This is also a collaborative study with the Inception study. Data for 600 patients will still need to be collected by the Inception study when our study starts. We will apply for our detailed questionnaires for 7 days (as per study 1A) to be administered to all the new patients that are included in the Inception study on a voluntary basis. This will allow us to capture data on almost 600 patients (150 of these will be from study 1A).

Using both our 150 studied patients from study1A and 450 patients in the Inception cohort (study 1B), we will then use cutting edge techniques in machine learning to ascertain if artificial intelligence (AI) can predict individuals who will develop chronic abdominal pain.

Study 2 and 3: Study 2 and 3 are a questionnaire-based cross-sectional study in patients with IBD (both CD and UC patients). The participants for study 2 are patients who are registered in IBD BOOST study and those for study 3 are patients who are registered in IBD BioResource (but not in IBD Boost study).

The aims are to determine the prevalence of chronic pain in Crohn's and UC patients, the prevalence of comorbid pain and IBS, lifestyle factors, and quality of life. IBD BOOST questionnaire is due to be administered to 10,000 patients. We will invite these patients to complete additional questionnaires not covered by IBD BOOST. We also approach 15,000 patients from IBD BioResourse who are not included in the IBD Boost study and administer questionnaires to them. We will be able to identify risk factors and aid a predictive model from static time point data if a number of those individuals have pain and a number do not. Further, in study 2 and 3, we will be able to determine whether the risk factors identified in study 1A and 1B accurately identify patients with and without chronic pain.

ELIGIBILITY:
Inclusion Criteria :

* Males or females who are over 18 years old.
* Patients who are diagnosed with UC or CD within 6 months before the enrolment.
* Patients who have access to the internet and have the IT skills to perform basic tasks e.g. operate emails and fill out questionnaires.
* Patients who are willing and able to participate in the study for the required duration, can understand and are willing to sign the consent forms and agree to undergo all protocol-related tests and procedures.

Exclusion Criteria:

* Patients who have severe extensive colitis and are at imminent risk of colectomy.
* Patients who already have the presence of a stoma or history of a fistula or stricture due to another diagnosis.
* Patients who are pregnant, lactating or thinking of becoming pregnant during the study period
* Patients who have unstable acute illness or exacerbation of an unstable chronic illness or chronic disease (other than IBD) that may affect assessments for this study as determined by previous physical examination, medical history, vital signs, ECG, and laboratory (serum biochemistry, hematology, urinalysis) assessments.
* Patients with a medical history of hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection that are not in remission and are on medication that can affect gastrointestinal function.
* Patients who have known or suspected to have a severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure (CHF) and chronic arrhythmia such as atrial fibrillation
* Patients who have known or suspected cerebrovascular disease (e.g. prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery)
* Patients who have a known history or suspected history of substance abuse or addiction (within the last five years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is males and females over the age of 18 who have been diagnosed with ulcerative colitis or Crohn's disease within the past 6 months before enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 25600 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of psychophysiological and biological risk factors for development of chronic abdominal pain | 3 years
  To identify psychophysiological and biological risk factors for the development of chronic abdominal pain in patients with newly diagnosed inflammatory bowel disease (ulcerative colitis and Crohn's disease) in a prospective longitudinal cohort study design
Build predictive models for chronic pain using artificial intelligence and machine learning | 3 years
  To use artificial intelligence (AI) and machine learning (ML) to build predictive models that use longitudinal data to identify patients who will develop chronic pain

SECONDARY OUTCOMES:
Chronic abdominal pain prevalence | 3 years
  To determine the prevalence of chronic abdominal pain
Co-morbid pain in IBD remission | 3 years
  To determine the prevalence of co-morbid pain in patients with IBD in remission
Lifestyle factors and quality of life | 3 years
  To study fatigue, lifestyle factors (e.g. sleep quality and dietary habits) and quality of life
Environmental sensitivity | 3 years
  To study environmental sensitivity in patients with IBD
Prevalence of IBS in IBD remission | 3 years
  To identify the prevalence of IBS in patients with IBD in remission

CONTACTS AND LOCATIONS:
Overall Officials: Qasim Aziz, Principal Investigator — Wingate Institute of Neurogastroenterology, Barts and the London School of Medicine and Dentistry, Queen Mary University of London
Locations (1):
- Neurogastroenterology, Barts and the London School of Medicine and Dentistry, Queen Mary University of London, London, United Kingdom